CLINICAL TRIAL: NCT03190161
Title: Music to Reduce Use of Smoking in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-00001
Record Dates: First submitted 2017-05-25; First posted 2017-06-16 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia; Nicotine Dependence; Smoking, Tobacco
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia; Tobacco Use Disorder; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Schizophrenia Patients (Experimental): Clinician verification diagnosis of Schizophrenia or Schizoaffective Disorder
  Interventions: Behavioral: Music session

INTERVENTIONS:
Behavioral: Music session — Participants will be asked to refrain from smoking from 24 hours before the music listening session as confirmed by breath carbon monoxide level <6 ppm on the day of the session. They will be contacted by phone or in person at the clinic as a reminder prior.

SUMMARY:
The purpose of this study is to explore the impact of self-selected music listening which targets disrupting the reward process maintaining smoking and additionally attenuating the reward processing deficits associated with schizophrenia. Five participants with schizophrenia/schizoaffective disorder who smoke/nicotine will participate in an individual session of self-selected music listening for a half an hour.

ELIGIBILITY:
Inclusion Criteria:

* clinician verification diagnosis of Schizophrenia or Schizoaffective Disorder
* smoked at least 10 cigarettes per day for the past month
* score of 4 or more on the Fagerstrom Test for Nicotine Dependence73
* psychiatric stability (e.g., no psychiatric hospitalizations within the last year, no expectation for medication change during study participation, no active suicidal ideation, no symptoms that interfere with ability to participate in study activities)
* the capacity to participate in the informed consent process

Exclusion Criteria:

* being medically unstable (e.g., medical condition that requires frequent medical appointments or hospitalizations and interferes with ability to participate in study activities)
* report active substance abuse or testing positive drug or alcohol use
* taking bupropion, varenicline, nicotine replacement products and/or involved in any other smoking cessation treatment
* participating in any treatment or activity that includes music as a focus
* having a seizure disorder, other neurological illnesses, or a family history of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Snaith-Hamilton Pleasure Scale (SHAPS) | 1 Day
  Measures Pleasure Pre Music Session
Snaith-Hamilton Pleasure Scale (SHAPS) Post Music Session | 1 Day
  Measures Pleasure Post Music Session
Pleasure Rating Scale (PRS) | 1 Day
  Measures Pleasure Pre Music Session
Pleasure Rating Scale (PRS) Post Music Session | 1 Day
  Measures Pleasure Post Music Session
Questionnaire of Smoking Urges-Brief (QSU-B) | 1 Day
  Measures Cravings Pre Music Session
Questionnaire of Smoking Urges-Brief (QSU-B) Post Music Session | 1 Day
  Measures Cravings Post Music Session
Minnesota Nicotine Withdrawal Scale (MNWS) | 1 Day
  Measures Withdrawal Pre Music Session and Post Music Session
Minnesota Nicotine Withdrawal Scale (MNWS) Post Music Session | 1 Day
  Measures Withdrawal Post Music Session

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Tracy, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States